CLINICAL TRIAL: NCT02755246
Title: Effect of Polyamine-enriched Dietary Supplementation on Cognitive Function in Healthy Older Adults With Subjective Cognitive Decline
Brief Title: Polyamine-enriched Diet in Healthy Older Adults With Subjective Cognitive Decline
Acronym: preSmartAge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Freie Universität Berlin, Institute of Biology/Genetic, Berlin,Germany (Unknown); Karl-Franzens-Universität Graz, Institute of Molecular Biosciences, Graz, Austria (Unknown)
Responsible Party: Principal Investigator, Claudia Schwarz, Postdoctoral Researcher, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: preSmartAge
Record Dates: First submitted 2016-04-05; First posted 2016-04-28 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Subjective Cognitive Decline
Keywords: subjective cognitive decline; dementia; lifestyle; polyamine; memory; elderly; prevention; treatment; dietary supplement; Polyamine-enriched diet
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Polyamine supplementation (Experimental): 750 mg polyamine-rich plant extract per day
  Interventions: Dietary Supplement: Polyamine supplementation
- Placebo (Placebo Comparator): 750 mg potato starch per day
  Interventions: Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: Polyamine supplementation — 3 months of polyamine supplementation (3 capsules/day)
  Arms: Polyamine supplementation
Dietary Supplement: Placebo supplementation — 3 months of placebo intake (3 capsules/day)
  Arms: Placebo

SUMMARY:
The overall objective of this study is to examine the effect of polyamine supplementation on cognitive performance of individuals with subjective cognitive decline.

DETAILED DESCRIPTION:
Memory abilities are known to decline during aging, a process that is accelerated in pathological conditions like subjective, mild cognitive impairment (MCI) and Alzheimer's disease (AD), all of which are a growing public-health concern with devastating effects. Polyamines supplementation and corresponding up-regulation of autophagy (i.e., cellular protein degradation pathways) may be a key target of intervention against age-related memory decline. The study will investigate whether a polyamine-enriched dietary supplementation (through capsule intake) could provide positive effects on the cognitive function of elderly individuals (60-80 years old) with subjective cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive healthy subjects with subjective memory decline and self-reported concerns
* 60-80 years old
* No manifest dementia (DSM-IV criteria)
* No limitations in activities of daily living
* Capacity for consent

Exclusion Criteria:

* Gluten, histamine or wheat seedling intolerance
* Severe neurological, internal or psychological diseases
* Advanced heart or respiratory diseases, severe arteriosclerosis, untreated thyroid disease or diabetes
* Malignant tumors, current or past history
* Brain tumors, stroke
* Disorders that impair attention
* Dementia
* Coagulation disorder, Marcumar or ASS therapy
* Drug abuse or alcohol dependency
* Current polyamine substitution

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function (from neuropsychological test battery) | Prior to intervention (baseline) and after 3 months of intervention
  Comparing changes in cognitive function in subjects with polyamine intake and placebo treatment (pre vs. post intervention)

SECONDARY OUTCOMES:
Laboratory parameters | Prior to intervention (baseline) and after 3 months of intervention
  comparing different markers derived from blood plasma like polyamine concentration (spermine, spermidine) and markers of inflammation pre vs. post intervention
Vascular parameters | Prior to intervention (baseline) and after 3 months of intervention
  Comparing intima-media-thickness pre vs. post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Background] Eisenberg T, Knauer H, Schauer A, Buttner S, Ruckenstuhl C, Carmona-Gutierrez D, Ring J, Schroeder S, Magnes C, Antonacci L, Fussi H, Deszcz L, Hartl R, Schraml E, Criollo A, Megalou E, Weiskopf D, Laun P, Heeren G, Breitenbach M, Grubeck-Loebenstein B, Herker E, Fahrenkrog B, Frohlich KU, Sinner F, Tavernarakis N, Minois N, Kroemer G, Madeo F. Induction of autophagy by spermidine promotes longevity. Nat Cell Biol. 2009 Nov;11(11):1305-14. doi: 10.1038/ncb1975. Epub 2009 Oct 4. PMID 19801973
- [Background] Gupta VK, Scheunemann L, Eisenberg T, Mertel S, Bhukel A, Koemans TS, Kramer JM, Liu KS, Schroeder S, Stunnenberg HG, Sinner F, Magnes C, Pieber TR, Dipt S, Fiala A, Schenck A, Schwaerzel M, Madeo F, Sigrist SJ. Restoring polyamines protects from age-induced memory impairment in an autophagy-dependent manner. Nat Neurosci. 2013 Oct;16(10):1453-60. doi: 10.1038/nn.3512. Epub 2013 Sep 1. PMID 23995066
- [Background] Ibe S, Kumada K, Yoshida K, Otobe K. Natto (fermented soybean) extract extends the adult lifespan of Caenorhabditis elegans. Biosci Biotechnol Biochem. 2013;77(2):392-4. doi: 10.1271/bbb.120726. Epub 2013 Feb 7. PMID 23391920
- [Background] Minois N, Carmona-Gutierrez D, Madeo F. Polyamines in aging and disease. Aging (Albany NY). 2011 Aug;3(8):716-32. doi: 10.18632/aging.100361. PMID 21869457
- [Background] Schaeffer V, Lavenir I, Ozcelik S, Tolnay M, Winkler DT, Goedert M. Stimulation of autophagy reduces neurodegeneration in a mouse model of human tauopathy. Brain. 2012 Jul;135(Pt 7):2169-77. doi: 10.1093/brain/aws143. Epub 2012 Jun 10. PMID 22689910
- [Background] Soda K, Dobashi Y, Kano Y, Tsujinaka S, Konishi F. Polyamine-rich food decreases age-associated pathology and mortality in aged mice. Exp Gerontol. 2009 Nov;44(11):727-32. doi: 10.1016/j.exger.2009.08.013. Epub 2009 Sep 6. PMID 19735716
- [Background] Soda K, Kano Y, Sakuragi M, Takao K, Lefor A, Konishi F. Long-term oral polyamine intake increases blood polyamine concentrations. J Nutr Sci Vitaminol (Tokyo). 2009 Aug;55(4):361-6. doi: 10.3177/jnsv.55.361. PMID 19763038
- [Background] Tiboldi A, Lentini A, Provenzano B, Tabolacci C, Hoger H, Beninati S, Lubec G. Hippocampal polyamine levels and transglutaminase activity are paralleling spatial memory retrieval in the C57BL/6J mouse. Hippocampus. 2012 May;22(5):1068-74. doi: 10.1002/hipo.22016. Epub 2012 Mar 30. PMID 22467251
- [Result] Wirth M, Benson G, Schwarz C, Kobe T, Grittner U, Schmitz D, Sigrist SJ, Bohlken J, Stekovic S, Madeo F, Floel A. The effect of spermidine on memory performance in older adults at risk for dementia: A randomized controlled trial. Cortex. 2018 Dec;109:181-188. doi: 10.1016/j.cortex.2018.09.014. Epub 2018 Oct 4. PMID 30388439
- [Result] Schwarz C, Stekovic S, Wirth M, Benson G, Royer P, Sigrist SJ, Pieber T, Dammbrueck C, Magnes C, Eisenberg T, Pendl T, Bohlken J, Kobe T, Madeo F, Floel A. Safety and tolerability of spermidine supplementation in mice and older adults with subjective cognitive decline. Aging (Albany NY). 2018 Jan 8;10(1):19-33. doi: 10.18632/aging.101354. PMID 29315079